CLINICAL TRIAL: NCT03365050
Title: Data Linkage Between NHS AAA Screening Programme and Primary Care Data to Determine the Safety of a Targeted Screening Programme.
Brief Title: A Study of the Safety of Targeted AAA Screening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0635
Record Dates: First submitted 2017-11-27; First posted 2017-12-07 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: AAA - Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention Given — No Intervention to be given

SUMMARY:
This study is a data linkage project within which we aim to model the impact on the NHS AAA Screening programme of a targeted approach to screening by targeting men who smoke. This in-silico study will generate a hypothetical population based on primary care datasets with known outcomes from screening (we know which men have an aneurysm and who do not) to determine the feasibility and safety of this approach.

DETAILED DESCRIPTION:
An abdominal aortic aneurysm (AAA) is present in 5-10% of men aged between 65 and 79 years and may be defined as an abdominal aortic diameter 3cm or above. In 2013 the NHS AAA screening programme (NAAASP) was fully rolled out across England with the aim of reducing AAA mortality in men aged 65 and over, based on evidence that screening reduces AAA-related mortality, and is highly cost effective. Within NAAASP, men with a large AAA (≤5.5cm) are referred for consideration of surgery whilst men with small AAA (≥5.4cm) are referred into surveillance (3.0-4.4cm: 1 year surveillance, 4.5-5.4cm: 3 months surveillance) as per standard operating procedures. In England 284,583 men were offered ultrasound screening (2015-2016), however, the number of men identified with AAA was 2,549 at a cost of approximately £7,755,000. This highlights one of the main problems with AAA screening in that the majority of men screened do not have disease. This also brought the number of men within AAA surveillance to 13,1047 whom do not require early surgery.

Several studies have investigated quality of life (QoL) in those who are screened for AAA, with one reporting short-term decreases in QoL at 1 year and four demonstrating no clinically important decrease in QoL in those screened positive compared with an unscreened control group. This has raised the issue of harms versus benefit however, AAA screening is not the same worldwide. For example, within The U.S. Preventive Services Task Force AAA Screening is recommended only for men aged 65-75 who have ever smoked as this group "stands to benefit the most from early detection and reparative surgical treatment due to a relatively higher prevalence of larger AAAs" . The screening programme described thus deemed men who have never smoked as lower risk for AAA and lower risk for rupture yet in England, we screen every man at the age of 65.

Although several risk factors for AAA have been identified, smoking is the only modifiable risk factor that has been associated with the development, expansion and rupture of AAA with a causative link revealed in vivo within a mouse model. Population based studies have also demonstrated that smoking prevalence over time is linked to changes in AAA mortality. It is possible that screening based on a history of smoking is feasible and safe, however, no evidence exists that this would be the case. In England details for men eligible for AAA screening is identified based on primary care data in that men registered with a General Practitioner (GP) who are 65 within that year are invited to screening. Primary care data may also be able to identify men with a history of smoking and other known risk factors for AAA including hypertension, heart disease and stroke.

ELIGIBILITY:
Inclusion Criteria:

* All men invited into the English AAA Screening Programme

Exclusion Criteria:

* All men not within the screening programme or who dissent from their data being used for research.

Ages: 65 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Men aged 65 who are invited for AAA screening in England.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
death from AAA after screening | long term mortality - 10 years
  AAA-related mortality after screening based on ONS ICD codes

SECONDARY OUTCOMES:
cost effectiveness analysis | long term - 10 years
  cost per QALY gained (cost-utility analysis) will be used to compare the current model of screening to a targeted model of screening as per NICE guidance.
Feasibility of targeted screening | 1 year
  Number of individuals identified with AAA in modelling study who have AAA at screening.
All-Cause mortality. | long term mortality - 10 years
  Death after screening based on ONS ICD codes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No